CLINICAL TRIAL: NCT01734720
Title: Common Bile Duct Stones - Natural History and Interventions : Data From the Swedish Registry for Gallstone Surgery and Endoscopic Retrograde Cholangio Pancreatography (ERCP) (GallRiks)
Brief Title: Common Bile Duct Stones - Natural History and Interventions
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Ersta Hospital, Sweden (Other)
Responsible Party: Principal Investigator, Mats Möller, MD. consultant suregon, Ersta Hospital, Karolinska Institutet
Other Study IDs: 2010/533-31/2
Record Dates: First submitted 2012-11-16; First posted 2012-11-28 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Common Bile Duct Stone
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- common bile duct stone: Patients undergoing cholecystectomy

SUMMARY:
The aims of this study were to

1. investigate what measures were taken when common bile duct stones (CBDS) were found intraoperatively in Sweden during the period May 2005 to December 2009 by using data from this population-based nationwide registry, and
2. analyze the outcome in terms of complications and success rates of bile duct clearance in relation to various stone sizes and interventions used. In order to further characterize the natural course of CBDS of various sizes, particular interest was focused on patients with positive findings where no peroperative measures to clear the bile ducts were taken or planned postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* common bile duct stones

Exclusion Criteria:

* none

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing cholecystectomy with common bile duct stones found in peroperative cholangiogram
Sampling Method: Non-Probability Sample
Enrollment: 3828 (Actual)
Dates: Start 2005-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
complications in relation to strategy for handling CBDS | 30 days post operative
  Complications reported to the registry at 30 day follow up after surgery

SECONDARY OUTCOMES:
complications in relation to stone size | 30 days post operative
  Complications reported to the registry at 30 day follow up after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mats Möller, MD, Principal Investigator — Karolinsks Institutet